CLINICAL TRIAL: NCT02287545
Title: Corneal Biomechanical Changes Following Trabeculectomy
Brief Title: Biomechanical Changes After Trabeculectomy
Acronym: TE-biomech
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Karin Pillunat, Medical Senior Doctor, Technische Universität Dresden
Other Study IDs: EK399122012
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Glaucoma, Primary
Keywords: open angle glaucoma; corneal biomechanics; trabeculectomy
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma, primary: Glaucoma patients undergoing trabeculectomy
  Interventions: Procedure: trabeculectomy

INTERVENTIONS:
Procedure: trabeculectomy — Standard trabeculectomy with the use of antimetabolites (mitomycin C) for glaucoma patients with insufficient intraocular pressure (IOP) control taking maximally tolerated IOP-reducing medication, visual field progression despite maximally tolerated IOP-reducing medication, adverse events because of maximally tolerated IOP-reducing medication or nono.compliance.
  Other Names: filtering glaucoma surgery

SUMMARY:
Corneal biomechanics are studied in glaucoma patients prior and at least 6 month after trabeculectomy.

DETAILED DESCRIPTION:
Prior to trabeculectomy corneal biomechanics are measured with the Ocular Response Analyzer (ORA, Reichert) and the Corvis st (Oculus). Both instruments work with an air-puff which deforms the cornea. Intraocular pressure is measured like in non-contact air-puff tonometry. The ORA also measures corneal hysteresis (CH) and the corneal resistance factor (CRF) which are qualitative measures of corneal biomechanics. The Corvis is a high-speed Scheimpflug-camera (4330 frames/sec) that records the quantitative movements of the cornea. At least 6 month after uncomplicated trabeculectomy the measurements are repeated.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patients in need of further IOP-reduction despite maximally tolerated therapy and assigned for trabeculectomy. Minimum of 18 years.

Exclusion Criteria:

* Corneal pathologies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary open-angle glaucoma patients assigened for a trabeculectomy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Corneal biomechanical changes following trabeculectomy | 2-3 years
  Evaluation of biomechanical properties of the cornea before and after trabeculectomy to evaluate whether intraocular pressure is accurately measured after trabeculectomy. Corneal hysteresis and corneal resistance factor as measured with the Ocular Response Analyzer and the corneal deformation response to an air-puff as measured with an ultra-high-speed Scheimpflug camera are assessed.

SECONDARY OUTCOMES:
Intraocular pressure after trabeculectomy | 2-3 years
  Intraocular pressure is measured with 3 different devices (Goldmann applanation tonometry, Ocular Response Analyzer, Corvis st) prior and at least 6 month after trabeculectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Karin R Pillunat, MD, Principal Investigator — Technische Universität Dresden
Locations (1):
- Technical University Dresden, Dresden, Saxony, Germany